CLINICAL TRIAL: NCT05991466
Title: The Effect of Dexmedetomidine on the Quality of Recovery in Parturients Undergoing Elective Caesarean Sections: a Randomized Comparative Study
Brief Title: Effect of Dexmedetomidine on the Quality of Recovery in Parturients Undergoing Elective Caesarean Sections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Youssef Ollaek, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MD-172-2021
Record Dates: First submitted 2023-06-26; First posted 2023-08-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-11

CONDITIONS: The Quality of Recovery (ObsQOR-11)
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group(A) (Active Comparator): Spinal anaesthesia will be performed with 0.5% hyperbaric bupivacaine 10-12 mg and TAP block will be performed with 30 ml 0.25% bupivacaine in each side.
  Interventions: Drug: Dexmedetomidine
- Group (B) (Active Comparator): Spinal anaesthesia will be performed with 0.5% hyperbaric bupivacaine10-12 mg and TAP block will be performed with 50 mcg Dexmedetomidine added to 30ml 0.25% bupivacaine in each side.
  Interventions: Drug: Dexmedetomidine
- Group (C) (Active Comparator): Spinal anaesthesia will be performed with 0.5% hyperbaric bupivacaine 10-12 mg added to 5 mcg dexmedetomidine. TAP block will be performed with 30ml 0.25% bupivacaine in each side.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — All patients will be assessed clinically and investigated for exclusion of any of the above-mentioned contraindications. The required laboratory work will be: complete blood count (CBC); prothrombin time and concentration (PT&PC); partial thromboplastin time (PTT); bleeding time (BT); clotting time (CT); liver function tests and kidney function tests.
  Before arrival to the operation room (OR), women will be premedicated by metoclopramide 10mg and ranitidine 50 mg intravenous. Intra operatively, hemodynamics will be recorded baseline before spinal anaesthesia , after its performance, every 3 minutes until delivery and then every 10 minutes till the end of the CS. Any change within 20% of baseline will be accepted and any changes more than 20% will be managed according to guidelines. All groups will be anaesthetized to preform CS with conventional spinal anaesthesia. The TAP block group will receive a landmark orientated Ultrasound guided bilateral TAP block.

SUMMARY:
The study hypothesizes that addition of dexmedetomidine to bupivacaine either in spinal anesthesia or TAP block is more effective and provide better ObsQor-11score than bupivacaine alone. Also, Dexmedetomidine in TAP block might provide a longer pain free time in comparison to intrathecal dexmedetomidine.

DETAILED DESCRIPTION:
Aim of the work To compare the quality of recovery (ObsQOR-11) in patients undergoing cesarean sections receiving dexmedetomedine either intrathecally or in the tap block in comparison to patients receiving conventional spinal anesthesia and tap block.

Statistical Analysis I. Sample size In a pilot study on 5 parturient who had undergone elective cesarean section under spinal anesthesia followed by TAP block with bupivacaine alone, the mean ObsQoR-11 at 24 hours was 65±9. In a single factor ANOVA study, sample size of 126 from the 3 groups is needed to detect a difference of at least 10 using the Tukey-Kramer (Pairwise) multiple comparison with study power of 83% and alpha error of 0.05. The common standard deviation within a group is assumed to be 9. The number of envelopes will be increased to 141 (47 per group) to compensate of possible 10% dropout. The sample size was calculated using PASS 15 Power Analysis and Sample Size Software (2017). NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass.

II. Statistical analysis Data will be coded and entered using the statistical package SPSS (statistical package for the social science) version 22. Data will be summarized using mean, standard deviation, median, minimum and maximum in quantitative data and using frequency (count) and relative frequency(percentage)for categorical data. Comparisons between quantitative variables will be done using the non parametric Mann-Whitney test. For comparing categorical data, Chi square (x2 ) test will be performed. Exact test will be used instead when the expected frequency is less than 5. P-value less than 0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be full-term pregnant females
* ASA classification I or ll.
* Aged between 18 and 40 years.
* Singleton pregnancy

Exclusion Criteria:

* Refusal of block.
* Bleeding disorders (platelets count <150,000; INR>1.5; PC<60%).
* wounds or infection at the puncture site.
* Known allergy to local anesthetic drugs.
* Contraindications to neuroaxial block.
* Contraindications to TAP block..

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of recovery score following CS (ObsQor-11) at the end of the first 24 hours postoperative. | 24 hours postoperative
  The mothers will be asked to rate each recovery item with an 11-point numerical Likert scale (0 = strongly negative; 10 = strongly positive).

SECONDARY OUTCOMES:
Time of first request of analgesia in hours | within 24 hours postoperative
  from time of spinal anesthesia to the first registration of VAS score more than 3
Ramsay sedation scale | 1, 2, 4, 6, 8, 12 and 24 hours
  1. Awake; agitated or restless or both
  2. Awake; cooperative, oriented, and tranquil
  3. Awake but responds to commands only
  4. Asleep; brisk response to light glabellar tap or loud auditory stimulus
  5. Asleep; sluggish response to light glabellar tap or loud auditory stimulus
  6. Asleep; no response to glabellar tap or loud auditory stimulus
Intra operative non-invasive mean blood pressure | within 24 hours postoperative
  in mmhg
Intra operative heart rate | within 24 hours postoperative
  beats per minutes
Visual Analogue Scale | 1, 2, 4, 6, 8, 12 and 24 hours postoperative
  VAS score at rest and during movement and cough The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Nausea and vomiting | intraoperative and postoperative 24 hours
  Nausea and vomiting
Onset of motor block using Bromage scale | Post spinal anesthesia up to 30 minutes
  defined as the time from giving spinal anesthesia until a modified Bromage score of IV will be reached),Duration of motor block (defined as the time from spinal anesthesia until Modified Bromage score of I).
Onset of sensory block | Post spinal anesthesia up to 30 minutes
  defined as the time needed to lose cold sensation when using the ice-cold test at the T6 dermatome level) and time to 2-segment regression of spinal anesthesia.
Neonatal Apgar score | at 1 and 5 minutes post delivery
  This scoring system provided a standardized assessment for infants after delivery. The Apgar score comprises five components: 1) color, 2) heart rate, 3) reflexes, 4) muscle tone, and 5) respiration, each of which is given a score of 0, 1, or 2.
Complications of spinal anaesthesia and TAP block | 12 hours post operative period.
  Complications of spinal anaesthesia and TAP block
Incidence of hypotension | post spinal anesthesia up to 1 hour
  systolic blood pressure < 90 or <70% of baseline
Incidence of bradycardia | post spinal anesthesia up to 1 hour
  heart rate less than 60 beats per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No